CLINICAL TRIAL: NCT04509128
Title: Echographic Characteristics of DIaphragm and FEmoral Quadriceps in COPD Patients: Evaluation of Their Relationship With the Lung Function Impairment and the Effect of Pulmonary Rehabilitation
Brief Title: Ultrasonographic Evaluation of Diaphragm and Quadriceps in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: EDIFEB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 19/19
Record Dates: First submitted 2020-08-03; First posted 2020-08-11 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: COPD; COPD Exacerbation
Keywords: Multidimensional evaluation; COPD; Pulmonary rehabilitation; Diaphragmatic ultrasound; Vastus lateralis muscle ultrasound
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- A: Subjects hospitalized for a COPD acute exacerbation, undergoing arterial blood gas analysis, evaluation of presence and grade of dyspnea, handgrip strength test, and diaphragmatic and vastus lateralis muscle ultrasound assessment, at admission and discharge.
- B: Subjects referred for pulmonary rehabilitation (PR) after a hospitalized COPD exacerbation, undergoing pulmonary function test, arterial blood gas analysis, evaluation of presence and grade of dyspnea, handgrip strength test, and diaphragmatic and vastus lateralis muscle ultrasound assessment, before and after PR.

SUMMARY:
The purpose of this study is to evaluate the prognostic role of echographic diaphragmatic assessment and vastus lateralis muscle ultrasound (US) in two independent populations of patients hospitalized for exacerbated Chronic Obstructive Pulmonary Disease (COPD) or undergoing pulmonary rehabilitation.

Specific aims of this protocol are: 1) to analyze the correlation between qualitative and quantitative US parameters and severity of illness indicators and respiratory function data; 2) to detect the postrehabilitation outcomes in terms of diaphragmatic and vastus lateralis muscle function, assessed by US, and the correlation between these outcomes and indicators of pulmonary rehabilitation treatment effectiveness; 3) to evaluate the ability of qualitative and quantitative US parameters to predict in-hospital mortality and length of stay; 4) to evaluate the ability of qualitative and quantitative US parameters to predict exacerbation rate, hospitalization rate and mortality rate six months after the discharge.

ELIGIBILITY:
Inclusion Criteria (Group A):

* COPD diagnosis
* previous or actual cigarette smoking history
* COPD exacerbation requiring hospitalization
* Obtained written informed consent

Exclusion Criteria:

* Pleural effusion extended for more than two intercostal spaces
* Interstitial lung diseases
* Major surgery in the previous 30 days
* Right pleurodesis or fibrothorax
* Right stroke outcomes
* Technical impossibility to perform ultrasound evaluations
* conditions, clinical or otherwise, that in the investigator's judgment may interfere with the study, or not recommending participation for security reasons
* Absence of written informed consent

Inclusion Criteria (Group B):

* COPD diagnosis
* previous or actual cigarette smoking history
* COPD exacerbation requiring hospitalization in the previous 30 days
* Indication to undergo a pulmonary rehabilitation protocol
* Obtained written informed consent

Exclusion Criteria:

* Pleural effusion extended for more than two intercostal spaces
* Interstitial lung diseases
* Major surgery in the previous 30 days
* Right pleurodesis or fibrothorax
* Right stroke outcomes
* Technical impossibility to perform ultrasound evaluations
* conditions, clinical or otherwise, that in the investigator's judgment may interfere with the study, or not recommending participation for security reasons
* Absence of written informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group A: Subjects hospitalizated for a COPD acute exacerbation Group B: Subjects referred for pulmonary rehabilitation (PR) after a hospitalized COPD exacerbation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Relationship between diaphragmatic and vastus lateralis muscle function and severity of illness indicators and respiratory function data | At discharge from hospital, estimated average of 10 days for Group A patients, and 28 days for Group B patients
  Evaluation of the correlation between qualitative and quantitative diaphragmatic and vastus lateralis muscle ultrasound parameters and the degree of respiratory function impairment
Variations of diaphragmatic and vastus lateralis muscle function, assessed by US, after 4 weeks of in-hospital Pulmonary Rehabilitation | After 4 weeks of Pulmonary Rehabilitation (T1)
  Evaluation of the post rehabilitation outcomes in terms of diaphragmatic and vastus lateralis muscle function
Relationship between post rehabilitation changes in diaphragmatic and vastus lateralis muscle function and indicators of pulmonary rehabilitation treatment effectiveness | After 4 weeks of Pulmonary Rehabilitation (T1)
  Evaluation of the correlation between post rehabilitation qualitative and quantitative diaphragmatic and vastus lateralis muscle ultrasound parameters and indicators of pulmonary rehabilitation treatment effectiveness (mMRC, Modified Medical Research Council, Dyspnea Scale; distance in meters at six minute walking test; respiratory function data; arterial blood gas values)

SECONDARY OUTCOMES:
Prediction of in-hospital mortality by means of parameters of diaphragmatic and vastus lateralis muscle function | At discharge from hospital, estimated average of 10 days for Group A patients, and 28 days for Group B patients
  Evaluation of the ability of qualitative and quantitative diaphragmatic and vastus lateralis muscle ultrasound parameters to predict in-hospital mortality
Prediction of length of stay by means of parameters of diaphragmatic and vastus lateralis muscle function | At discharge from hospital, estimated average of 10 days for Group A patients, and 28 days for Group B patients
  Evaluation of the ability of qualitative and quantitative diaphragmatic and vastus lateralis muscle ultrasound parameters to predict length of stay
Prediction of COPD exacerbation rate by means of parameters of diaphragmatic and vastus lateralis muscle function | Six months after discharge (T2)
  Evaluation the ability of qualitative and quantitative US parameters to predict COPD exacerbation rate six months after the discharge
Prediction of hospitalization rate by means of parameters of diaphragmatic and vastus lateralis muscle function | Six months after discharge (T2)
  Evaluation the ability of qualitative and quantitative US parameters to predict hospitalization rate six months after the discharge
Prediction of mortality rate by means of parameters of diaphragmatic and vastus lateralis muscle function | Six months after discharge (T2)
  Evaluation the ability of qualitative and quantitative US parameters to predict mortality rate six months after the discharge

CONTACTS AND LOCATIONS:
Overall Officials: Vittoria Conti, PhD, Principal Investigator — Unit of Pulmonay Rehabilitation, IRCCS San Raffaele Pisana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Decramer M, De Benedetto F, Del Ponte A, Marinari S. Systemic effects of COPD. Respir Med. 2005 Dec;99 Suppl B:S3-10. doi: 10.1016/j.rmed.2005.09.010. Epub 2005 Oct 10. PMID 16219454
- [Background] Koerts-de Lang E, Schols AM, Rooyackers OE, Gayan-Ramirez G, Decramer M, Wouters EF. Different effects of corticosteroid-induced muscle wasting compared with undernutrition on rat diaphragm energy metabolism. Eur J Appl Physiol. 2000 Aug;82(5-6):493-8. doi: 10.1007/s004210000231. PMID 10985606
- [Background] Decramer M, Lacquet LM, Fagard R, Rogiers P. Corticosteroids contribute to muscle weakness in chronic airflow obstruction. Am J Respir Crit Care Med. 1994 Jul;150(1):11-6. doi: 10.1164/ajrccm.150.1.8025735.
- [Background] Sabino PG, Silva BM, Brunetto AF. Nutritional status is related to fat-free mass, exercise capacity and inspiratory strength in severe chronic obstructive pulmonary disease patients. Clinics (Sao Paulo). 2010 Jun;65(6):599-605. doi: 10.1590/S1807-59322010000600007. PMID 20613936
- [Background] Marquis K, Debigare R, Lacasse Y, LeBlanc P, Jobin J, Carrier G, Maltais F. Midthigh muscle cross-sectional area is a better predictor of mortality than body mass index in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2002 Sep 15;166(6):809-13. doi: 10.1164/rccm.2107031. PMID 12231489
- [Background] Montes de Oca M, Torres SH, Gonzalez Y, Romero E, Hernandez N, Mata A, Talamo C. Peripheral muscle composition and health status in patients with COPD. Respir Med. 2006 Oct;100(10):1800-6. doi: 10.1016/j.rmed.2006.01.020. Epub 2006 Mar 20. PMID 16545558
- [Background] Thurlbeck WM. Diaphragm and body weight in emphysema. Thorax. 1978 Aug;33(4):483-7. doi: 10.1136/thx.33.4.483. PMID 694801
- [Background] Arora NS, Rochester DF. Effect of body weight and muscularity on human diaphragm muscle mass, thickness, and area. J Appl Physiol Respir Environ Exerc Physiol. 1982 Jan;52(1):64-70. doi: 10.1152/jappl.1982.52.1.64. PMID 7061279
- [Background] Rochester DF. The diaphragm: contractile properties and fatigue. J Clin Invest. 1985 May;75(5):1397-402. doi: 10.1172/JCI111841. No abstract available. PMID 3889054
- [Background] Cesari M, Pedone C, Chiurco D, Cortese L, Conte ME, Scarlata S, Incalzi RA. Physical performance, sarcopenia and respiratory function in older patients with chronic obstructive pulmonary disease. Age Ageing. 2012 Mar;41(2):237-41. doi: 10.1093/ageing/afr167. Epub 2011 Dec 8. No abstract available. PMID 22156558
- [Background] Ticinesi A, Meschi T, Narici MV, Lauretani F, Maggio M. Muscle Ultrasound and Sarcopenia in Older Individuals: A Clinical Perspective. J Am Med Dir Assoc. 2017 Apr 1;18(4):290-300. doi: 10.1016/j.jamda.2016.11.013. Epub 2017 Feb 13. PMID 28202349
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] McLean RR, Shardell MD, Alley DE, Cawthon PM, Fragala MS, Harris TB, Kenny AM, Peters KW, Ferrucci L, Guralnik JM, Kritchevsky SB, Kiel DP, Vassileva MT, Xue QL, Perera S, Studenski SA, Dam TT. Criteria for clinically relevant weakness and low lean mass and their longitudinal association with incident mobility impairment and mortality: the foundation for the National Institutes of Health (FNIH) sarcopenia project. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):576-83. doi: 10.1093/gerona/glu012. PMID 24737560
- [Background] Cesari M, Landi F, Calvani R, Cherubini A, Di Bari M, Kortebein P, Del Signore S, Le Lain R, Vellas B, Pahor M, Roubenoff R, Bernabei R, Marzetti E; SPRINTT Consortium. Rationale for a preliminary operational definition of physical frailty and sarcopenia in the SPRINTT trial. Aging Clin Exp Res. 2017 Feb;29(1):81-88. doi: 10.1007/s40520-016-0716-1. Epub 2017 Feb 10. PMID 28188558
- [Background] Ticinesi A, Narici MV, Lauretani F, Nouvenne A, Colizzi E, Mantovani M, Corsonello A, Landi F, Meschi T, Maggio M. Assessing sarcopenia with vastus lateralis muscle ultrasound: an operative protocol. Aging Clin Exp Res. 2018 Dec;30(12):1437-1443. doi: 10.1007/s40520-018-0958-1. Epub 2018 Apr 26. PMID 29700758
- [Background] Iwasawa T, Takahashi H, Ogura T, Asakura A, Gotoh T, Shibata H, Inoue T. Influence of the distribution of emphysema on diaphragmatic motion in patients with chronic obstructive pulmonary disease. Jpn J Radiol. 2011 May;29(4):256-64. doi: 10.1007/s11604-010-0552-8. Epub 2011 May 24. PMID 21607839
- [Background] Podnar S, Harlander M. Phrenic nerve conduction studies in patients with chronic obstructive pulmonary disease. Muscle Nerve. 2013 Apr;47(4):504-9. doi: 10.1002/mus.23617. Epub 2013 Feb 4. PMID 23382059
- [Background] Zanforlin A, Giannuzzi R, Nardini S, Testa A, Soldati G, Copetti R, Marchetti G, Valente S, Inchingolo R, Smargiassi A. The role of chest ultrasonography in the management of respiratory diseases: document I. Multidiscip Respir Med. 2013 Aug 9;8(1):54. doi: 10.1186/2049-6958-8-54. PMID 23937880
- [Background] Rodrigues FM, Demeyer H, Loeckx M, Hornikx M, Van Remoortel H, Janssens W, Troosters T. Health status deterioration in subjects with mild to moderate airflow obstruction, a six years observational study. Respir Res. 2019 May 18;20(1):93. doi: 10.1186/s12931-019-1061-7. PMID 31103027
- [Background] Martinez CH, Diaz AA, Meldrum CA, McDonald MN, Murray S, Kinney GL, Hokanson JE, Curtis JL, Bowler RP, Han MK, Washko GR, Regan EA; COPDGene Investigators. Handgrip Strength in Chronic Obstructive Pulmonary Disease. Associations with Acute Exacerbations and Body Composition. Ann Am Thorac Soc. 2017 Nov;14(11):1638-1645. doi: 10.1513/AnnalsATS.201610-821OC. PMID 29090990
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Crimi C, Heffler E, Augelletti T, Campisi R, Noto A, Vancheri C, Crimi N. Utility of ultrasound assessment of diaphragmatic function before and after pulmonary rehabilitation in COPD patients. Int J Chron Obstruct Pulmon Dis. 2018 Oct 8;13:3131-3139. doi: 10.2147/COPD.S171134. eCollection 2018. PMID 30349221
- [Background] Bolton CE, Bevan-Smith EF, Blakey JD, Crowe P, Elkin SL, Garrod R, Greening NJ, Heslop K, Hull JH, Man WD, Morgan MD, Proud D, Roberts CM, Sewell L, Singh SJ, Walker PP, Walmsley S; British Thoracic Society Pulmonary Rehabilitation Guideline Development Group; British Thoracic Society Standards of Care Committee. British Thoracic Society guideline on pulmonary rehabilitation in adults. Thorax. 2013 Sep;68 Suppl 2:ii1-30. doi: 10.1136/thoraxjnl-2013-203808. No abstract available. PMID 23880483
- [Background] Singanayagam A, Schembri S, Chalmers JD. Predictors of mortality in hospitalized adults with acute exacerbation of chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2013 Apr;10(2):81-9. doi: 10.1513/AnnalsATS.201208-043OC. PMID 23607835
- [Background] Scarlata S, Mancini D, Laudisio A, Benigni A, Antonelli Incalzi R. Reproducibility and Clinical Correlates of Supine Diaphragmatic Motion Measured by M-Mode Ultrasonography in Healthy Volunteers. Respiration. 2018;96(3):259-266. doi: 10.1159/000489229. Epub 2018 Aug 16. PMID 30114702
- [Background] Scarlata S, Mancini D, Laudisio A, Raffaele AI. Reproducibility of diaphragmatic thickness measured by M-mode ultrasonography in healthy volunteers. Respir Physiol Neurobiol. 2019 Feb;260:58-62. doi: 10.1016/j.resp.2018.12.004. Epub 2018 Dec 13. PMID 30553945
- See also: GOLD (Global Initiative for Chronic Obstructive Lung Disease) guidelines — https://goldcopd.org/wp-content/uploads/2018/11/GOLD-2019-v1.7-FINAL-14Nov2018-WMS.pdf